CLINICAL TRIAL: NCT04524533
Title: Delivery of a Smoking Cessation Induction Intervention Via Virtual Reality (VR) Headset During a Dental Cleaning: Randomized Controlled Trial
Brief Title: VR Smoking Cessation During a Dental Hygiene Visit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: H-40368; 4UH3DE028866-02 (NIH)
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
Keywords: video-based smoking cessation; smoking cessation evidence-based treatments (EBTs); text messages; dental cleaning; smoking cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research assistants who are collecting outcome data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized into the intervention arm will watch smoking cessation videos (ready to quit or not ready to quit) during a dental cleaning clinic visit, receive a brochure about EBTs, and participate in a 4-week text message program which consists of automated and tailored text messages to motivate EBT utilization. After the 4-week program, the intervention group will receive monthly assessment text messages.
  Interventions: Behavioral: Experimental smoking cessation video; Other: Brochure of smoking cessation EBTs; Behavioral: Tailored text message program
- Control group (Active Comparator): Participants randomized into the control arm will watch a control video during a dental hygiene visit and receive a brochure about EBTs, and a 4-week assessment-only text message program.
  Interventions: Behavioral: Control video; Other: Brochure of smoking cessation EBTs; Other: Assessment text messages

INTERVENTIONS:
Behavioral: Experimental smoking cessation video — Participants who are randomized to the intervention group will watch an educational video that includes tips on quitting smoking during a dental cleaning. The video is approximately 10 minutes long and tailored to readiness to quit at the time of the dental visit.
  Arms: Intervention group
Behavioral: Control video — Participants randomized to the control group will watch a 10 minute video.
  Arms: Control group
Other: Brochure of smoking cessation EBTs — All participants will receive identical print materials on EBTs consistent with smoking cessation standard clinical care.
Behavioral: Tailored text message program — Participants randomized to the intervention group will be enrolled in a 4-week tailored text message program which includes assessment questions in addition to text messages geared towards motivating and facilitating EBT utilization for individuals ready to quit smoking and individuals who are not ready to quit smoking.
  Arms: Intervention group
Other: Assessment text messages — Participants randomized to the control group will be enrolled in a different 4-week text message program that includes only assessment questions.
  Arms: Control group

SUMMARY:
The goal of this randomized controlled trial (RCT) is to test whether a smoking cessation induction intervention delivered during a dental cleaning appointment increases the utilization of evidence-based treatments (EBTs) for smoking cessation within 7 months post-dental cleaning appointment.

Approximately 400 cigarette smokers who are scheduled for a dental cleaning appointment at the Boston University Goldman School of Dental Medicine (BUGSDM) patient treatment center will be recruited and enrolled. Participants will be randomized to either the intervention or control group

DETAILED DESCRIPTION:
Approximately 400 patients who have a scheduled prophylaxis, root planing and scaling dental appointment at the BUGSDM patient treatment center will be recruited and enrolled in the randomized controlled trial. Participants who complete the baseline survey will be randomized to either the intervention or control group. The intervention group will watch one of two smoking cessation videos during the appointment (depending on readiness to quit), receive a brochure about EBTs for smoking cessation, and participate in a 4-week tailored text message program designed to motivate EBT utilization. After the 4-week text message program, the intervention group will receive monthly assessment text messages for six months. The control group will watch a control video during the appointment, receive the same brochure about EBTs as the intervention group, and participate in an assessment-only 4-week text message program. All videos are approximately 10 minutes long.

After the dental clinic appointment, all participants will complete an online questionnaire and begin the 4-week text message program.

At the end of the 4-week text message program, and 3 and 6 months later, all participants will complete online questionnaires.

Primary Aim 1: To test the efficacy of the intervention vs. control in increasing utilization of EBTs over the course of follow-up (7-months). Hypothesis 1.1: Smokers randomized to the intervention will be more likely to engage with (contact) EBTs. Hypothesis 1.2: Smokers randomized to the intervention will have greater treatment utilization (e.g., more days in the text message program, more days using smoking cessation medication, and more quitline counseling sessions, greater number of EBTs).

Secondary Aims:

Aim 2: To test the effect of the intervention vs. controls on quit attempts and on motivation to quit. Hypothesis 2: Smokers randomized to the intervention will have more quit attempts and higher motivation to quit.

Aim 3: To test the efficacy of the intervention vs controls on biochemically verified abstinence. Hypothesis 3: Smokers randomized to the intervention will have higher quit rates at follow-up.

Aim 4: To assess the mechanisms through which the intervention effects occur (social cognitive mediators) and to identify subpopulations for whom intervention effects differ (moderators, e.g., readiness to quit, gender, race/ethnicity). Hypothesis 4: The intervention will directly affect the putative mediators, which will in turn affect EBT utilization. The role of moderators will be exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the Boston University, Henry M Goldman School of Dental Medicine treatment center with an upcoming dental hygiene appointment (dental prophylaxis or scaling and root planing)
* Self-reported smoking 100 cigarettes or more (not including e-cigarettes or vaping) in lifetime
* Self-reported smoking any cigarette (not including e-cigarettes or vaping) in the preceding week
* Self-reported cigarettes (not including e-cigarettes or vaping) 'some days', 'most days' or 'every day' in the preceding week
* Is able to understand written and spoken study materials
* Score of 'Never,' 'Rarely' or 'Sometimes' on the validated single-item literacy screener ("How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor, dentist, or pharmacy?")
* Self-reported visual capacity to watch a video as indicated by the score 'Some difficulty' or 'No difficulty' to: "How much difficulty do you have with your vision, even when wearing glasses?"
* Self-reported ability to wear headphones that are inserted partially inside the ear
* Self-reported use of text messaging at least once in the preceding month
* Self-reported access to necessary resources for intervention: Cell phone capable of text messaging
* Live in Massachusetts
* Stated willingness to comply with text message program procedures (receive and respond to text messages for 4-weeks)

Exclusion Criteria:

* Participation in another treatment or intervention study for smoking cessation or research involving text messaging
* Current use of medications for smoking cessation or smoking reduction (nicotine replacement product, or non-nicotine medications) whether prescribed or not
* Failure to complete the pre-dental clinic appointment procedure before the start of the dental appointment (opt-into the text message program and complete the baseline questionnaire)
* Failure to show up to scheduled dental appointment at the clinic
* Previous participation in the pilot phase
* Could not watch video during dental appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Utilization of Massachusetts State Quitline | 7 months
  Self-reported use of smoker quitline services validated through objective review of the quitline database (whether participant contacted the quitline, whether a decision to start counseling was made, the type of counseling requested, the number of sessions received, whether a quit date was set, whether nicotine replacement products were requested by participants, and whether nicotine replacement products were sent to participants).
Utilization of the National Cancer Institute "SmokefreeTXT" service | 7 months
  Self-reported use of SmokefreeTXT validated through objective verification of program interaction (length of program utilization, and engagement with program).
Utilization of clinic or hospital-based smoking cessation services | 7 months
  Self-reported use of smoking cessation programs offered by clinics or hospitals (whether participant contacted the clinic, whether a decision to start counseling was made, the type of counseling requested, the number of sessions received, whether a quit date was set, whether nicotine replacement products and/or other cessation medications were requested by participants, and whether nicotine replacement products and/or other cessation medications were given to participants).

SECONDARY OUTCOMES:
Use of a combination of EBTs | 7 months
  Self-reported use of at least two EBTs for smoking cessation validated through objective verification of program use.
Quit smoking attempts | 7 months
  Self-reported number of quit smoking attempts lasting 24 hours or more.
Motivation to quit smoking | 7 months
  Self-reported motivation to quit smoking within the following 30 days.
7-day point prevalence smoking abstinence at end-of-treatment | 1 month
  Self-reported smoking abstinence biochemically confirmed with cotinine test.
7-day point prevalence smoking abstinence at end-of-treatment | 3 months
  Self-reported smoking abstinence biochemically confirmed with cotinine test.
7-day point prevalence smoking abstinence at end-of-treatment | 6 months
  Self-reported smoking abstinence biochemically confirmed with cotinine test.
Participant's satisfaction | within 10 days after the dental clinic visit.
  Self-reported satisfaction with overall experience at the dental clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Borrelli, PhD, Principal Investigator — Henry M Goldman School of Dental Medicine
Locations (1):
- Henry M Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
To enable verification of outcome measures, participant's data will be shared with the smoker quitline service and with the industry partner managing the text message programs.

REFERENCES:
- [Derived] Hart NJ, Goodman MS, Park H, Endrighi R, Jurasic MM, Cabral HJ, Borrelli B. Factors associated with dental fear and anxiety among smokers in urban dental clinics: a cross-sectional analysis. BMC Oral Health. 2026 Jan 13. doi: 10.1186/s12903-026-07682-3. Online ahead of print. PMID 41526906
- [Derived] Borrelli B, Endrighi R, Jurasic MM, Hernandez H, Jones E, Ospina J, Cabral HJ, Quintiliani LM, Werntz S. A smoking cessation induction intervention via virtual reality headset during a dental cleaning: protocol for a randomized controlled trial. BMC Public Health. 2022 May 31;22(1):1074. doi: 10.1186/s12889-022-13427-y. PMID 35641925

DOCUMENTS (1):
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT04524533/ICF_000.pdf